CLINICAL TRIAL: NCT04777266
Title: The Music Therapy for People With Schizophrenia and Relates Psychosis: Effects on Symptoms, Self-esteem, Self-stigma, Social Cognition, Social Functioning and Quality of Live. Clinical Trial.
Brief Title: Music Therapy for People With Schizophrenia and Relates Psychosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State reference center for psychosocial care (Other Government)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Sergio Lacamara Cano, Psychologist, State reference center for psychosocial care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StateReferenceCenter
Record Dates: First submitted 2021-02-05; First posted 2021-03-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Psychosis
Keywords: Music Therapy; Psychosis; Adjunct Therapy; Psychosocial Rehabilitation; Recovery
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Music Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Music therapy Group (Experimental): experimental group receiving the MT programme in addition to their usual treatment (pharmacological and psychosocial) (TAU + MT)
  Interventions: Behavioral: Music therapy and treatment as usual
- Control Non music therapy group (Active Comparator): Group with usual treatment only (TAU).
  Interventions: Behavioral: Music therapy and treatment as usual

INTERVENTIONS:
Behavioral: Music therapy and treatment as usual — The session-based intervention programme was designed with an integrated and multimodal perspective of music therapy [37], which allows the combination of active and passive activities together with focuses and perspectives based on empirical evidence [38]. It was implemented using a process-based approach, adapting content to different phases in the process: initial contact, managing resistance, confidence building, relationships, awareness, and closure. The central focus is on the patient and to adapt and remain flexible in the sessions in accordance with the capabilities and needs of the group members. Different perspectives are integrated via nonverbal communication. The layout and any changes to the setting are made in a gradual way in keeping with the process to foster feelings of security and belonging. Sessions begin with a brief period of breathing which then moves into warming-up and free-expression using instruments, followed by the central activity and the closure.

SUMMARY:
Treatment of symptoms, rehabilitation of cognitive deficits, improvement of social functioning and quality of life in schizophrenia and other psychoses are approached through a comprehensive strategy that combines psychopharmacology with psychosocial interventions. However, despite the efficacy of these interventions, this is not the same in all patients, and a large percentage do not achieve functional recovery.

DETAILED DESCRIPTION:
The aim of this research is to carry out a randomized trial on the effects of a music therapy (MT) program, implemented in addition to the usual pharmacological and psychosocial rehabilitation (TAU), on symptoms, self-esteem, internalized stigma, social cognition, social functioning and the quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be diagnosed with schizophrenia or schizoaffective disorder in accordance with DSM-IV-TR criteria using the Structured Clinical Interview for DSM-IV-TR (SCID-I).
* The patients will all clinically stable with a diagnosis of schizophrenia and regularly attended in the state approved centre for psychosocial attention CREAP (Centro de Referencia Estatal para la Atención Psicosocial) in Valencia (Spain).

Exclusion Criteria:

* Previous brain damage
* Substance abuse in the last year
* Display of mood disorders
* Organic or substance based mental disorders
* Disrupted symptomatology
* Serious symptoms with difficulty in understanding the implications of informed consent and not replying in the interviews and assessment questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 10 weeks
  Symptoms of schizophrenia are measured according to the subscale scores and total score on the PANSS which consists of 30 items scored from 1 (Absent) to 7 (Extreme). Scores range from 30 to 210, with higher scores indicating more symptoms.
State-Trait Anxiety Inventory (STAI) | 10 weeks
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic.Scores range from 20 to 80, with higher scores correlating with greater anxiety.
World Health Organization Quality of Life-Short version (WHOQOL-BREF) | 10 weeks
  The WHOQOL-BREF contains 24 questions covering 4 domains plus two questions related to overall quality of life and satisfaction with health. Highes scores represent higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sergio Lacamara Cano, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided